CLINICAL TRIAL: NCT02056366
Title: The Effect of α-lipoic Acid Treatment in Patient With Cardiac Autonomic Neuropathy by Comparing the Change of HRV Index & ANS Function:A 6month Multicenter, Randomized, Open Label Clinical Trial CANON Study
Brief Title: The Effect of α-lipoic Acid Treatment in Patient With Cardiac Autonomic Neuropathy
Acronym: CANON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Chong Hwa Kim, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALA_IIT01
Record Dates: First submitted 2014-02-03; First posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes; Cardiac Autonomic Neuropathy
Keywords: Cardiac Autonomic Neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- α-lipoic acid (Active Comparator): α-lipoic acid PO medication, 600mg per day, for 6weeks α-lipoic acid PO medication, 1200mg per day, for 6weeks
  Interventions: Drug: α-lipoic acid
- No treatment group (No Intervention): No Intervention

INTERVENTIONS:
Drug: α-lipoic acid — α-lipoic acid 600mg PO medication,Per day, For 6weeks α-lipoic acid 1200mg PO medication,Per day, For 6weeks
  Other Names: Neuropaid OD Tablet
  Arms: α-lipoic acid

SUMMARY:
The purpose of this study is to see if it is safe and effective to give alpha lipoic acid in people with cardiac autonomic neuropathy(CAN). Cardiac autonomic neuropathy(CAN) affects the nerves that control heart rate and blood flow to the heart in people with diabetes. CAN may cause problems with the rhythm of the heartbeat or decrease blood flow to the heart.

DETAILED DESCRIPTION:
Study type : Interventional Study Design : Allocation: Randomized Control: no treatment Endpoint Classification: Safety/Efficacy Study Intervention Model: Parallel Assignment Masking: Open Label Primary Purpose: Treatment Primary Outcome Measures : Heart rate variability(HRV) Index

Secondary Outcome Measures : Autonomic Nerve System(ANS) function 5 test, EuroQoL 5-Dimension Questionnaire(EQ-5D)

ELIGIBILITY:
Inclusion Criteria :

* Established Cardiac Autonomic Neuropathy in type 2 diabetes.
* aged 20 years to 80 years
* Capable of giving informed consent

Exclusion Criteria :

* History of other significant disease such as the nerve system (Parkinson's disease, epilepsy, multiple sclerosis), hepatic disease, hypothyroid, etc Other medical condition or treatment likely to affect the autonomic nerve system
* HbA1C > 11%
* Not controlled hypertension (SBP≥160mmHg, DBP≥100mmHg)
* Diagnosed ketoacidosis within 4 weeks
* Unstable cardiac disease (unstable angina or myocardial infarction )
* Pregnancy
* Involvement in other clinical trial in last 4 weeks
* Known or suspected sensitivity to trial products

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy of α-lipoic Acid in patients with cardiac autonomic neuropathy | up to 24weeks
  check the Heart rate variability(HRV) Index

SECONDARY OUTCOMES:
Secondary Efficacy of α-lipoic Acid in patients with cardiac autonomic neuropathy | up to 24weeks
  Check the Autonomic Nerve System(ANS) function 5 test

OTHER OUTCOMES:
Number of Patients with Adverse events as a Measure of Safety | up to 24weeks
  Check the Number of Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bong Yun Cha, MD, PhD, Principal Investigator — The Catholic University of Korea
Locations (3):
- South Korea (3):
  - The Catholic University of Korea, Seoul, Seoul
  - Eulji General Hospital, Seoul, Seoul
  - Sejong General Hospital, Seoul, Seoul